CLINICAL TRIAL: NCT03534882
Title: Prospective, Randomized, Single-blind Controlled Trial of Topical Prostaglandin Analogue Washout Following Chronic Monotherapy in Adults With Suspected or Proper Primary Open Angle Glaucoma
Brief Title: Effects of Prostaglandin Analogue Washout Following Long-term Therapy in Adults With Primary Open Angle Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cindy Hutnik (Other)
Responsible Party: Sponsor-Investigator, Cindy Hutnik, Ophthalmology, Glaucoma Specialist, Western University, Canada
Organization: Western University, Canada (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4834
Record Dates: First submitted 2018-05-11; First posted 2018-05-23 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Primary Open-Angle Glaucoma, Mild Stage; Glaucoma, Suspect; Ocular Hypertension
Keywords: anti-glaucoma medications; glaucoma; prostaglandin analogues; medication washout
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma

STUDY DESIGN:
Intervention Model Description: This randomized-controlled trial studies patients with primary open angle glaucoma or ocular hypertension currently treated with topical IOP-lowering prostaglandin analogue (PGA) medications. Patients meeting inclusion criteria and having none of the exclusion criteria are contacted. If interested, patients meet research staff to discuss the study protocol and informed consent is obtained. Participants are randomized to one of two groups (A or B). Allocation to group is concealed to physicians. Participants have their IOP measured at Day 0. Group A patients are asked to discontinue their PGA for 42 days. Group B patients continue their medications as prescribed by their physician. Patients are closely followed, where IOP is measured on day 7, 21, and 42 in all participants. Once the assessment is complete, participants are debriefed on the nature of the study and potential findings. At the end of trial, participants resume standard therapy according to CJO 2009 Glaucoma Guidelines.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Washout (Experimental): Discontinuation of topical prostaglandin analogue therapy: Participants are asked to discontinue (washout) their prostaglandin analogue for 42 days. As the experimental group, the purpose of this arm is to determine the lingering IOP-reducing effects following discontinuation of chronic prostaglandin analogue therapy, and to determine if IOP rises back to baseline (pre-treatment values).
  Interventions: Other: Discontinuation of topical prostaglandin analogue therapy
- Control (No Intervention): Patients are asked to remain on their prostaglandin analogues and continue treatment as prescribed by their ophthalmologist. The purpose of this arm is to minimize bias in intraocular pressure readings.

INTERVENTIONS:
Other: Discontinuation of topical prostaglandin analogue therapy — Participants are asked to discontinue their prostaglandin analogue eye drops for the designated time period (42 days)
  Other Names: Medication washout
  Arms: Washout

SUMMARY:
A target for glaucoma treatment is the intra-ocular pressure (IOP) which is lowered with medications, laser, or surgical intervention. The efficacy of different medication classes is well understood as their IOP lowering effects have been well documented. However, beyond the basic biochemical and pharmacokinetic actions, long-term effects of these drugs on IOP have not been adequately studied. Specifically, does long-term use of anti-glaucoma medications have lasting effects on IOP even with subsequent discontinuation of the medication? In Ontario, prostaglandin analogues are the most frequently prescribed first line anti-glaucoma medication. In our study, we examine the lingering IOP-reducing effects of the prostaglandin analogue anti-glaucoma drug class. Our overall objective is to determine if patients previously treated with prostaglandin analogues remain within acceptable treatment ranges 6 weeks after medication discontinuation, and if this IOP differs from pre-treatment baseline values. Half of participants will discontinue their prostaglandin analogue (PGA) treatment for 6 weeks, while the other half will continue their PGA therapy as prescribed by their ophthalmologist. Both groups will be followed closely throughout the 6 weeks to monitor changes in IOP. This can help us understand the lasting effects of medication use and can help better guide clinical care in optimizing glaucoma management, and help direct study designs of future research that involve any therapy secondary to prostaglandin analogue treatment.

DETAILED DESCRIPTION:
Quality assurance plan: Paper copies of all registry data is securely stored at the site of data collection. Registry data is first de-identified and then stored in an encrypted Master data excel sheet that only research staff have access to.

Data Checks and Source Data Verification: Data is monitored closely and re-assessed frequently by multiple members of the research team to ensure the accuracy of the Master data excel sheet. Registry data will be compared to paper registry copies and patient medical records to ensure accuracy and completeness.

Standard Operating Procedures:

All patients currently being seen by Dr. Hutnik (~6000) will have their charts reviewed. Personal information will be recorded to allow research staff to contact eligible participants. Clinical information recorded includes: diagnosis, intraocular pressure (IOP) at baseline, IOP at subsequent follow up visits with medication use, medication history, surgical and laser intervention history, visual acuity at baseline and follow-up visits, and visual field mean deviation. Patients fulfilling the inclusion and having none of the exclusion criteria are contacted via telephone by the research staff to invite them to participate in the trial. If they are interested, participants are met with in-person and provided with an information package including a form of consent. Research staff provide detailed description of this study's protocol, risks, and benefits for the patient prior to obtaining informed consent. Patients are also provided with the research teams' contact information should they have any questions or concerns. As part of the information package, participants receive notice that should they experience worrisome signs and symptoms, they should contact their ophthalmologist's office immediately. Following enrolment, participants are given an enveloped that randomizes them two either the control group (continues their eye drop medications) or experimental group (temporarily discontinues eye drop medications). In order to eliminate measurement bias, this allocation is concealed to research staff until completion of the trial. Participants' IOP is measured by Goldmann applanation tonometry at day of allocation (Day 0) and subsequently 7, 21, and 42 days after. In addition, should their IOP increase back to baseline levels prior to their final day of pressure measurement, participants are asked to restart their eye drops and are closely followed to ensure their IOPs return back to their pre-study values. Paper copies of participant signed consent and information form are stored in the research database. Once the assessment is complete, all participants will be debriefed on the nature of the study and potential findings. At the end of trial, participants will resume standard therapy according to Canadian Ophthalmology Society (COS) 2009 Glaucoma Guidelines.

Power analysis using a General Linear Multivariate Model for Power and Sample Size (GLIMMPSE) found that a total patient N value of 87 (154 eyes) was sufficient power for our study

Missing Data: All missing data is documented in the Master data record and will be reported. Participants with missing baseline (pre-treatment) IOP values are excluded from the study. Within-study missing IOP values are accounted for in statistical analysis.

Statistical analysis: Statistical analysis is performed on R. Data is analyzed using a linear mixed effects model fit by restricted maximum likelihood (REML) t-tests with Satterthwaite approximations to compare mean intraocular pressure between control and washout groups at day 0, 7, 21, and 42.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of glaucoma or or ocular hypertension
* Prostaglandin analogue responder >20% intraocular pressure (IOP) reduction from baseline
* Age >18 years
* Baseline IOP (pre-treatment) ≥21 mmHg
* Prostaglandin analogue treatment duration > 6 months

Exclusion Criteria:

* Diagnosis of acute angle closure glaucoma
* Treatment with > 1 glaucoma medication
* Topical steroid > 3 consecutive weeks
* Intraocular surgery in last 6 months prior to enrollment
* Glaucoma laser intervention in last 12 months prior to enrollment
* Best Corrected Visual Acuity (BCVA) < 70 letters (EDTRS or Snellen equivalent)
* Visual field mean deviation <-3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2014-05-27 (Actual); Primary Completion 2017-06-22 (Actual); Study Completion 2017-06-22 (Actual)

PRIMARY OUTCOMES:
Day 42 Intraocular Pressure (mmHg) | 42 days after starting trial
  Measured by Goldmann Applanation Tonometer

SECONDARY OUTCOMES:
Day 7 Intraocular Pressure (mmHg) | 7 days after starting trial
  Measured by Goldmann Applanation Tonometer
Day 21 Intraocular Pressure (mmHg) | 21 days after starting trial
  Measured by Goldmann Applanation Tonometer

CONTACTS AND LOCATIONS:
Overall Officials: Cindy ML Hutnik, MD, PhD, Principal Investigator — Western University, Department of Ophthalmology
Locations (1):
- Ivey Eye Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kass MA, Heuer DK, Higginbotham EJ, Johnson CA, Keltner JL, Miller JP, Parrish RK 2nd, Wilson MR, Gordon MO. The Ocular Hypertension Treatment Study: a randomized trial determines that topical ocular hypotensive medication delays or prevents the onset of primary open-angle glaucoma. Arch Ophthalmol. 2002 Jun;120(6):701-13; discussion 829-30. doi: 10.1001/archopht.120.6.701. PMID 12049574
- [Background] Tataru CP, Purcarea VL. Antiglaucoma pharmacotherapy. J Med Life. 2012 Sep 15;5(3):247-51. Epub 2012 Sep 25. PMID 23049625
- [Background] Lee R, Hutnik CM. Projected cost comparison of selective laser trabeculoplasty versus glaucoma medication in the Ontario Health Insurance Plan. Can J Ophthalmol. 2006 Aug;41(4):449-56. doi: 10.1016/S0008-4182(06)80006-2. PMID 16883360
- [Background] Kreidler SM, Muller KE, Grunwald GK, Ringham BM, Coker-Dukowitz ZT, Sakhadeo UR, Baron AE, Glueck DH. GLIMMPSE: Online Power Computation for Linear Models with and without a Baseline Covariate. J Stat Softw. 2013 Sep;54(10):i10. doi: 10.18637/jss.v054.i10. PMID 24403868
- [Derived] Lim CW, Diaconita V, Liu E, Ault N, Lizotte D, Nguyen M, Hutnik CML. Effect of 6-week washout period on intraocular pressure following chronic prostaglandin analogue treatment: a randomized controlled trial. Can J Ophthalmol. 2020 Apr;55(2):143-151. doi: 10.1016/j.jcjo.2019.08.004. Epub 2019 Nov 8. PMID 31712013